CLINICAL TRIAL: NCT01579812
Title: A Phase II Evaluation of Metformin, Targeting Cancer Stem Cells for the Prevention of Relapse in Patients With Stage IIC/III/IV Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: Evaluation of Metformin, Targeting Cancer Stem Cells for Prevention of Relapse in Gynecologic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2011.037; HUM 47900 (Other: Univ Mich Medical School Institutional Review Board (IRBMED))
Record Dates: First submitted 2012-03-30; First posted 2012-04-18 (Estimated); Results first posted 2018-05-25 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Keywords: Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Patients receiving primary surgical debulking followed by adjuvant chemotherapy will initiate metformin prior to primary surgery. Following surgery patients will be initiated on metformin prior to the initiation of chemotherapy.
  Patients treated with neoadjuvant chemotherapy will be initiated on metformin prior to the initiation of chemotherapy. Following surgery patients will be initiated on metformin prior to the re-initiation of chemotherapy.
  Other Names: Fortamet, Glucophage, Glumetza, Riomet

SUMMARY:
The primary objective of this study is to determine if metformin administered in combination with chemotherapy to women with advanced ovarian, primary peritoneal or fallopian tube cancer will improve recurrence-free survival at 18 months compared to controls.

DETAILED DESCRIPTION:
Despite 70% remission rates with surgery and chemotherapy, the majority of patients with stage III/IV ovarian cancer will relapse and die of their disease. This is consistent with a cancer stem cell (CSC) model in which a few residual treatment resistant stem cells persist and initiate disease recurrence. Laboratory studies indicate therapies targeting CSC will greatly improve cancer outcomes. We have recently characterized a population of CSC in ovarian cancer. Importantly, similar to that observed in breast cancer, we have found that the diabetes drug metformin can restrict ovarian CSC growth and proliferation. In addition metformin increases tumor cell sensitivity to chemotherapy. Consistent with this, epidemiologic studies demonstrate that diabetic patients with ovarian cancer taking metformin have better outcomes than those not taking metformin. However, metformin has not been tested as an anti-cancer stem cell agent in ovarian cancer. Thus we propose to perform a phase II clinical trial using metformin as an anti-cancer stem cell agent in ovarian cancer patients. Patients who plan to receive primary surgical debulking will initiate metformin therapy prior to surgery and then continue after surgery along with chemotherapy. Patients who will be treated neoadjuvantly will initiate metformin with chemotherapy prior to surgery and then continue both metformin and chemotherapy after surgery. Tumor specimens will be acquired for all patients at the time of primary surgery. The primary objective of this study will be to determine if metformin improves the recurrence-free survival (RFS) of patients relative to historical controls. Secondary objectives of this study will be: (a) to compare the amount of CSC in primary tumor specimens in metformin treated patients versus matched controls from our tumor bank, (b) to determine if metformin improves overall survival relative to historical controls, (c) to confirm the safety of metformin in non-diabetic ovarian cancer patients, and (d) as laboratory studies indicate that metformin is most active in p53 mutant cells and p53 is mutated in ~50% of ovarian cancers, we will assess whether response rates correlate with p53 mutation status. If successful, this well tolerated FDA approved drug could be immediately translated into phase III trials and impact patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with potential diagnosis of ovarian, fallopian, or primary peritoneal cancer.
2. Care plan including surgical debulking and traditional adjuvant or neo-adjuvant chemotherapy (6-9 cycles of platinum and taxane based therapy).
3. Eastern Cooperative Oncology Group performance status 0-2.
4. Age > 18 years or < 80 years.
5. Adequate renal function (serum creatinine <1.4mg/dL).
6. Adequate liver function (bilirubin < 1.5 times ULN).

   * Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) < 5 times the upper limit of normal in case of liver metastases.
   * ALT or AST < 2.5 times the ULN in absence of liver metastases.
7. Ability to understand and complete written informed consent.
8. Mentally, physically, and geographically able to undergo treatment and follow up.

Exclusion Criteria:

1. Patients diabetes mellitus. (Patients with only a history of gestational diabetes will be allowed to be included in the study.)
2. Metformin use in the last 6 months.
3. A known hypersensitivity to metformin.
4. A history of metabolic acidosis, including ketoacidosis or increased risk of lactic acidosis.
5. Pregnancy or Lactation.
6. Patients who have any severe and/or uncontrolled medical conditions.
7. Patients with a history of renal disease.
8. Patients with other known active malignancy (excluding adequately treated basal cell / squamous cell skin cancer, in situ cancer, or other cancer for which the patient has been disease free for 2 years).
9. Patients receiving any other investigational agents.

Ages: 19 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-10; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J. Buckanovich, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Brown JR, Chan DK, Shank JJ, Griffith KA, Fan H, Szulawski R, Yang K, Reynolds RK, Johnston C, McLean K, Uppal S, Liu JR, Cabrera L, Taylor SE, Orr BC, Modugno F, Mehta P, Bregenzer M, Mehta G, Shen H, Coffman LG, Buckanovich RJ. Phase II clinical trial of metformin as a cancer stem cell-targeting agent in ovarian cancer. JCI Insight. 2020 Jun 4;5(11):e133247. doi: 10.1172/jci.insight.133247. PMID 32369446

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin
Started | 90
Completed | 38
Not Completed | 52
Not completed — Ineligible after treatment start | 40
Not completed — Patient choice | 3
Not completed — Noncompliance | 3
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 90
Age, Continuous [Mean (Full Range); unit: years] | 58 [30 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 69
  Unknown or Not Reported | 19

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-Free Survival
Description: Determine the percentage of patients alive without recurrence at 18 months. Investigators will also determine recurrence free survival when patients with persistent disease are excluded.
  Definition of progression or recurrence and survival will be defined as increasing clinical, radiological or histological evidence of disease since study entry or two serum values of CA-125 greater than or equal to two times the upper limits of normal (ULN) performed at least one week apart, regardless of CT scan results.
  Recurrence-Free Interval will be defined as date from start of chemotherapy to the date of first clinical, biochemical, or radiological evidence of progression or death due to any cause.
Time Frame: 18 months
Population: 90 patients were enrolled, only 38 completed treatment and were analyzed. Patients found to have persistent disease were censored at the time they were found to have progressive disease. 11 patients had persistent disease.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Metformin - All Patients Analyzed: Metformin: Patients receiving primary surgical debulking followed by adjuvant chemotherapy will initiate metformin prior to primary surgery. Following surgery patients will be initiated on metformin prior to the initiation of chemotherapy.
  Patients treated with neoadjuvant chemotherapy will be initiated on metformin prior to the initiation of chemotherapy. Following surgery patients will be initiated on metformin prior to the re-initiation of chemotherapy.
- Metformin - Patients With Persistent Disease Excluded: Metformin: Patients receiving primary surgical debulking followed by adjuvant chemotherapy will initiate metformin prior to primary surgery. Following surgery patients will be initiated on metformin prior to the initiation of chemotherapy.
  Patients treated with neoadjuvant chemotherapy will be initiated on metformin prior to the initiation of chemotherapy. Following surgery patients will be initiated on metformin prior to the re-initiation of chemotherapy.
  Patients with persistent disease were excluded in this analysis.
Arm/Group | Metformin - All Patients Analyzed | Metformin - Patients With Persistent Disease Excluded
Number analyzed (Participants) | 38 | 27
percentage of patients | 58.1 [38 to 73.8] | 55.6 [35.2 to 71.8]

2. Secondary Outcome: Overall Survival
Description: Determine the median overall survival time for all patients who complete treatment as well as for patients presenting with stage IIc/ III and stage IV ovarian cancer.
Time Frame: Up to 3 Years
Population: 90 patients were enrolled and only 38 patients completed treatment. 25 of the 38 patients had stage IIc/III ovarian cancer. 13 of the 38 patients had stage IV ovarian cancer.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Metformin - Patients Stage IIc/ III Ovarian Cancer: Patients with stage IIc/ III ovarian cancer receiving primary surgical debulking followed by adjuvant chemotherapy will initiate metformin prior to primary surgery. Following surgery patients will be initiated on metformin prior to the initiation of chemotherapy.
- Metformin - Patients With Stage IV Ovarian Cancer: Patients with stage IV ovarian cancer receiving primary surgical debulking followed by adjuvant chemotherapy will initiate metformin prior to primary surgery. Following surgery patients will be initiated on metformin prior to the initiation of chemotherapy.
Arm/Group | Metformin - All Patients Analyzed | Metformin - Patients Stage IIc/ III Ovarian Cancer | Metformin - Patients With Stage IV Ovarian Cancer
Number analyzed (Participants) | 38 | 25 | 13
months | 43 [35 to 56] | 52 [35 to 65] | 36 [15 to 43]

ADVERSE EVENTS:
Time Frame: Up to 30 days post treatment
Arm/Group | Metformin
All-Cause Mortality (participants affected / at risk) | 2/90
Serious Adverse Events (participants affected / at risk) | 26/90
Other Adverse Events (participants affected / at risk) | 40/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=90)
Anemia (Blood and lymphatic system disorders) | 6 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Asystole (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 6 (6)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 4 (4)
White blood cell decreased (Investigations) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=90)
Anemia (Blood and lymphatic system disorders) | 26 (70)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 13 (19)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 12 (13)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 17 (21)
Fever (General disorders) | 2 (2)
Infusion related reaction (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 4 (5)
Allergic reaction (Immune system disorders) | 1 (1)
Nail infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (7)
Alkaline phosphatase increased (Investigations) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 8 (10)
Creatinine increased (Investigations) | 4 (4)
Lymphocyte count decreased (Investigations) | 1 (2)
Neutrophil count decreased (Investigations) | 12 (17)
Platelet count decreased (Investigations) | 13 (28)
Weight loss (Investigations) | 4 (4)
White blood cell decreased (Investigations) | 17 (34)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (10)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 6 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 5 (9)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Concentration impairment (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4)
Headache (Nervous system disorders) | 3 (3)
Paresthesia (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 6 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (10)
Anxiety (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 3 (3)
Restlessness (Psychiatric disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (4)
Hot flashes (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT01579812/Prot_SAP_000.pdf